CLINICAL TRIAL: NCT02324413
Title: Randomised Controlled Pilot Study: Does Intraoperative Clonidine Reduce the Incidence of Post-hospitalisation Negative Behaviour Changes in Children Who Are Distressed During the Induction of General Anaesthesia?
Brief Title: Pilot Study: Intraoperative Clonidine and Postoperative Behaviour
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Richard Beringer (Other)
Responsible Party: Sponsor-Investigator, Richard Beringer, Dr, University Hospitals Bristol and Weston NHS Foundation Trust
Organization: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CH-2011-3668
Record Dates: First submitted 2014-01-16; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Negative Behaviour Change
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clonidine (Active Comparator): Clonidine intravenous 1 or 2 micrograms / kg
  Interventions: Drug: Clonidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — Comparison between placebo and 2 different concentrations of clonidine
  Arms: clonidine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Children who are upset during induction of general anaesthesia are frequently distressed postoperatively and are more likely to demonstrate negative behaviour changes.

This pilot study is a randomised controlled study of clonidine vs placebo during anaesthesia to identify whether postoperative behavioural disturbance may be minimised.

ELIGIBILITY:
Inclusion Criteria:

* age 2 to 10 years inclusive
* healthy (ASA 1 or 2)

Exclusion Criteria:

* inability of parents to understand english

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of negative changes on the post-hospitalization behavior questionnaire | 24 hours and 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol Dental Hospital, Bristol, United Kingdom